CLINICAL TRIAL: NCT05626244
Title: Ser Pai & Ser Mãe: Avaliação de Uma intervenção Parental Para crianças Com Problemas
Brief Title: Being a Parent: Evaluation of a Parenting Intervention for Childhood Behavioral Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida (Other)
Collaborators: Fundação Cecília Zino (Unknown); King's College London (Other)
Responsible Party: Principal Investigator, Laura Maciel, Ph.D. Student, ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EPEC_PT_2020
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Childhood Behavior Problems; Positive Parenting Skills; Parental Concerns; Parents' Sense of Competence
Keywords: Parenting Interventions; Childhood; Behavior Problems; Positve Parenting
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial will have two arms, namely the intervention group and the waitlist control group.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will be receiving the parenting intervention (name of the intervention: Being a Parent).
  Interventions: Behavioral: Being a Parent
- Waitlist Control Group (No Intervention): The control group will be in a waitilist condition, in which they will not receive any intervention during the trial, but posteriorly will have the opportunity to receive the parenting intervention.

INTERVENTIONS:
Behavioral: Being a Parent — Being a Parent (BaP) is a group parenting intervention for parents of children (2-11 years old) with behavioral problems. It consists of 2-hour sessions facilitated by psychologists for between 8-12 parents. Based on attachment, family systems, and cognitive-behavioral theories, BaP successfully integrates knowledge acquisition, behavior change with adult learning and social support. Each course session is highly interactive involving an engaging blend of small and large group discussion, role play, demonstrations, information sharing and reflection. This enables parents to practice and use new skills to achieve specific goals (Day et al., 2020).
  Arms: Intervention Group

SUMMARY:
This randomized controlled trial aims to test the efficacy of an early parenting intervention for childhood behavior problems in the portuguese community. More specifically, this research intends to: 1) examine the effects of the parenting intervention in childhood behavior problems, positive parenting skills and parental concerns; 2) test participants' adherence, acceptability and dropout rates of the parenting intervention; and 3) qualitatively analyze the experience of parents' who received the intervention.

Researchers will compare an intervention group with a waitlist control group to see if there are any significant differences between these groups regarding childhood behavior problems and the aforementioned parenting dimensions.

Participants in both groups will be able to participate in the parenting intervention that has a duration of 9 weeks. Furthermore, they will be asked to fill in pre and post data.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregivers who identify difficulties managing the behavior of a child between the ages of 2 and 11 years old.

Exclusion Criteria:

* Primary caregivers of children with serious neurodevelopmental or cognitive disorders diagnosed;
* Primary caregivers of children institucionalized;
* Primary caregivers who do not comprehend, read or write in portuguese;
* Primary caregivers inability to commit to weekly sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-09 (Actual); Study Completion 2023-12-09 (Actual)

PRIMARY OUTCOMES:
Change in the Child Behavior Checklist for Preschool and School Years (CBCL; Achenbach & Rescorla, 2001; Portuguese version: Achenbach et al., 2014) | Through study completion, up to 11 months
  Based on parents' reports, it assesses behaviors that have been present for the past six months in youth between the ages of 1.5 and 18 years old. Each item is assessed using a 3-point Likert scale, ranging from Not True to Completely True. Only the broadband Externalizing Domain and its subdimensions will be used, which assesses behavioral problems, and comprises 28 items for the Preschool Years and 71 for the School Years.

SECONDARY OUTCOMES:
Change in the Parental Concerns Scale (Castro, 2012) | Through study completion, up to 11 months
  It is constituted by 21 items, divided into five concern dimensions, namely family and school problems; eating, sleep and physical complaints; preparation; fears; and negative behaviors. Parents must answer using a 5-point Likert scale (Not concerned to Extremely concerned).
Change in the Parental Sense of Competence (PSOC; Johnston & Mash, 1989; portuguese version: Nunes et al., 2014) | Through study completion, up to 11 months
  Measures parental sense of competence as perceived by parents, by examining two dimensions, namely Efficacy and Satisfaction.
Change in the Parental Styles and Dimensions Questionnaire (PSDQ; Robinson et al., 2001; portuguese version: Pedro et al., 2015) | Through study completion, up to 11 months
  Analyzes dysfunctional parenting practices.

OTHER OUTCOMES:
Research Qualitative Interview | Through study completion, up to 11 months
  Qualitative interviews will be carried out with a selection of parents who received the parenting intervnetion in order to analyze they experience and overall satisfaction of the parenting intervention

CONTACTS AND LOCATIONS:
Overall Officials: Laura Maciel, Ph.D. student, Principal Investigator — Ispa - Instituto Universitário
Locations (1):
- Ispa - Instituto Universitário, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maciel L, Basto-Pereira M, Day C. Reducing childhood externalizing behavior: A feasibility RCT of the being a Parent program. Behav Res Ther. 2025 Jun;189:104737. doi: 10.1016/j.brat.2025.104737. Epub 2025 Apr 1. PMID 40239337